CLINICAL TRIAL: NCT01216540
Title: Occurrence and Economic Impact of Nephrotoxicity Associated With Vancomycin Exposure
Brief Title: Vancomycin-Associated Nephrotoxicity
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Principal Investigator, Vanessa Stevens, Principal Investigator, University at Buffalo
Other Study IDs: IIS-000184
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Nephrotoxicity
Keywords: vancomycin; nephrotoxicity; length of stay; costs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving vancomycin

SUMMARY:
The primary goal of this study is to determine if there is an association between greater exposure to vancomycin and the development of nephrotoxicity. The secondary goal is to estimate the costs to the hospital associated with these nephrotoxic events.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at time of hospital admission
* Had an absolute neutrophil count of ≥ 1000 cells/mm^3
* Received > 48 hours of intravenous vancomycin therapy
* Had one or more vancomycin trough levels reported within the 96 hours after therapy initiation
* Had a baseline serum creatinine level of < 2.0 mg/dL and baseline creatinine clearance level of ≥ 30 mL/min

Exclusion Criteria:

* Previous diagnosis of cystic fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A simple random sample of 400 patients treated with greater than 48 hours of intravenous vancomycin exposure during hospitalization during the time period from July 1, 2009 through June 30, 2010
Sampling Method: Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2010-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Time to nephrotoxicity | within 72 hours post completion of vancomycin therapy

SECONDARY OUTCOMES:
Hospital costs | until discharge
Length of stay | until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jack Brown, PharmD, Principal Investigator — State University of New York at Buffalo; Vanessa Stevens, PhD, Principal Investigator — Internal Medicine, Division of Epidemiology, University of Utah School of Medicine
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States